CLINICAL TRIAL: NCT01840904
Title: Subjective Sleep Quality and Fatigue During and After Acute Uncomplicated Diverticulitis
Brief Title: Subjective Sleep and Fatigue During and After Acute Diverticulitis
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Ismail Gögenür, Senior resident and D.Sc., Herlev Hospital
Other Study IDs: CHU-3
Record Dates: First submitted 2013-04-13; First posted 2013-04-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Acute Diverticulitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute uncomplicated diverticulitis: CT-verified acute uncomplicated diverticulitis managed by antibiotics

SUMMARY:
The purpose of this study is to investigate subjective sleep quality and fatigue during and after Acute uncomplicated diverticulitis assessed by questionnaires and a sleep-diary. The investigators hypothesis is that subjective sleep and fatigue are correlated with the inflammatory activities.

DETAILED DESCRIPTION:
An increasing number of experimental studies have showed that inflammation can induce disturbances in sleep architecture, mediated by cytokines. some studies showed that cytokines also induce daytime fatigue. In this study the investigators aim to describe the patient experiences of sleep and fatigue during the acute inflammation and the recovery, and the investigators seek to exam the correlation of fatigue with Polysomnography-measured night sleep and cytokine levels in plasma.

Following methods will be applied

* Other: Karolinska Sleepiness Scale
* Other: Physical Fatigue Scale
* Other: Visual Analog Scale and 10 point-scales to measure fatigue, general well-being, subjective sleep and pain
* Other: Sleep-diary
* Device: Polysomnograph - Embla Titanium (Natus Medical Incorporated, USA)
* Procedure: Plasma cytokines (IL-2, IL-6 and TNF-alfa(tumor necrosis factor))
* Procedure: Plasma CRP(C reactive protein) and leukocytes
* Device: Wrist-Actigraph - Octagonal Basic Motionlogger, Ambulatory monitoring Inc, New York, USA

ELIGIBILITY:
Inclusion Criteria:

* CT-verified diverticulitis patients managed by antibiotic treatment at Herlev Hospital
* Pain and fever occurred less than 72 hours prior to the admission
* ASA (American Society of Anesthesiologists) score I to III

Exclusion Criteria:

* Surgical intervention needed
* Complicated diverticulitis
* Complications in relation to diverticulitis
* Pain and fever occurred more than 72 hours prior to the admission
* In anticoagulant treatment and heart rate control treatment
* Known Autoimmune disease
* Known medically treated sleep-disorder (insomnia, restless legs etc.) and sleep apnea
* Shift-work or jetlag
* Daily use of opioid, psychopharmaca, opioids or anxiolytics (including Hypnotics)
* Known psychiatry conditions in treatment with psychopharmaca
* Daily alcohol intake of more than 5 units or drug abuse
* Missing written consent
* Diabetes Mellitus
* Predicted bad compliance
* Pregnant or breast-feeding
* Urine or fecal incontinence
* Severe kidney disease
* Current cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 x Acute uncomplicated diverticulitis (Hansen and stock stage 1) patients aged 18-75 years managed by antibiotic treatment at Herlev Hospital.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Changes in Sleep quality during acute uncomplicated diverticulitis from baseline score at remission (14th, 21st and 30th day) | 1st-10th day and 14th, 21st, 30th day following the admission
  1. subjective sleep quality measured by a Visual Analog Scale (VAS) at given time frame
  2. sleep-diary recording sleep quantity of day and night sleep at given time frame
Changes in Sleepiness during acute uncomplicated diverticulitis from baseline score at remission (14th, 21st and 30th day) | 1st-10th day and 14th, 21st, 30th day following the admission
  Sleepiness measured by Karolinska Sleepiness Scale at given time frame
Changes in fatigue during acute uncomplicated diverticulitis from baseline score at remission (14th, 21st and 30th day) | 1st-10th day and 14th, 21st, 30th day following the admission
  1. General fatigue measured on Visual Analog Scale at given time frame
  2. Physical fatigue measured on a 10 points scale at given time frame
Changes in general well-being during acute uncomplicated diverticulitis from baseline score at remission (14th, 21st and 30th day) | 1st-10th day and 14th, 21st, 30th day following the admission
  general well being measured on VAS
Changes in pain during acute uncomplicated diverticulitis from baseline score at remission (14th, 21st and 30th day) | 1st-10th day and 14th, 21st, 30th day following the admission
  Pain measured on VAS

SECONDARY OUTCOMES:
accuracy of sleep diary compared to actigraph in measuring sleep data | 1st-10th day and 14th, 21st, 30th day following the admission
  Sleep quantity registered by the sleep diary compared with actigraph measured sleep quantity at given time frame
accuracy of sleep diary compared to Polysomnography (PSG) in measuring sleep data | 1st-2nd day and 30th day following the admission
  Sleep quantity registered by the sleep diary compared with PSG measured sleep quantity at given time frame
correlation between fatigue and level of cytokines in patient's plasma | 1st and 2nd and 30th day following the admission
  Investigator seek to find correlations between levels of IL-2, IL-6, TNF-alpha, CRP, Leucocytes and subjective fatigue measured by VAS and a 10 points scale.
correlation between pain and level of cytokines in patient's plasma | 1st and 2nd and 30th day following the admission
  Investigator seek to find correlations between levels of IL-2, IL-6, TNF-alpha, CRP, Leucocytes and subjective pain measured by VAS.
correlation between sleepiness and level of cytokines in patient's plasma | 1st and 2nd and 30th day following the admission
  Investigator seek to find correlations between levels of IL-2, IL-6, TNF-alpha, CRP, Leucocytes and subjective sleepiness measured by Karolinsk Sleepiness Scale
correlation between general well-being and level of cytokines in patient's plasma | 1st and 2nd and 30th day following the admission
  Investigator seek to find correlations between levels of IL-2, IL-6, TNF-alpha, CRP, Leucocytes and general well-being measured by VAS

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, M.D., Principal Investigator — University of Copenhagen, Herlev Hospital
Locations (1):
- Department D, Herlev Hospital, Herlev, Copenhagen, Denmark